CLINICAL TRIAL: NCT04233944
Title: Effectiveness of Integrated Livelihood and Nutrition Interventions to Improve Maternal and Child Nutrition and Health in Rural Uganda: A Birth Cohort Study
Brief Title: Uganda Birth Cohort Study
Acronym: UBC
Status: Terminated | Type: Observational
Why Stopped: Funding constraints
Sponsor: Tufts University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Makerere University (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Patrick Webb, Program Director, Tufts University
Other Study IDs: 11302
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Birth Outcomes; Stunting; Wasting; Anemia
Keywords: Birth Outcomes; Pregnancy; Aflatoxin; Environmental Enteric Dysfunction (EED); Growth; Stunting; Wasting; Uganda; Anemia
MeSH Terms: conditions — Growth Disorders; Cachexia; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women and their infants: Mothers and their infants were followed throughout the first two years of the infant's life. Data were collected at enrollment, birth, 3, 6, 9,12, 18 and 24 months from the date of delivery.

SUMMARY:
The UBC was a USAID-funded longitudinal prospective cohort study of pregnant women (n= 5030) aged 15-49 years from rural North and South-Western regions of Uganda, conducted between 2014 and 2016. The aim of the UBC study was to observationally follow pregnant women and their newborns until 2 years of age and compare changes over time in communities that were part of an ongoing USAID project called the Community Connector (CC) compared to those communities that were not included in the Community Connector project.

DETAILED DESCRIPTION:
This study aimed to assess the role of livelihoods, agriculture and nutrition in improving maternal and child nutrition and health in rural Uganda in communities that were a part of an ongoing program that was un-related to the study. The overall aim of this study was to understand the effect of participating in an ongoing program that provided support on nutrition, agriculture, water, hygiene and sanitation and the change over time in the nutritional status of mothers and children under two years of age. The specific objectives of this observational study were as follows:

1. To compare health and nutrition status of pregnant women in communities participating in the Community Connector project to those that were not participating in the program
2. To assess the aflatoxin levels in pregnancy and test its association with birth outcomes and early life growth as measured by weight and length
3. To assess environmental enteropathy in pregnancy and test its association with birth outcomes and early life growth
4. To assess access to coverage and adherence to information/messages and engagement in Community Connector project's activities
5. To determine heterogeneity in program exposure and variability in household and agro-ecological characteristics and its relationship with maternal and infant health and nutrition status

ELIGIBILITY:
Inclusion criteria:

Inclusion into pregnancy surveillance:

* Participant is a woman aged 15-49 years
* Participant intends to reside in the study area through the enrollment period
* Participant provides informed consent herself or through a legal guardian

Inclusion into main study:

* Pregnancy is confirmed by urine pregnancy test
* Mother is aged 15-49 years
* Mother intends to reside in the study area through completion of follow-up
* Mother intends to deliver in the study area
* Mother provides informed consent (potentially as an emancipated minor)

Exclusion criteria:

-None

Ages: 15 Years to 49 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Pregnant women, children under two years, and their households in Northern and Southwestern Uganda during 2014-2016
Sampling Method: Probability Sample
Enrollment: 5044 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
Percent of infants who were stunted | 0-2 years old
  Percent of infants with a height-for-age less than -2 standard deviations
Percent of infants who were wasted | 0-2 years old
  Percent of infants with a weight-for-height less than -2 standard deviations
Percent of infants who were underweight | 0-2 years old
  Percent of infants with a weight-for-age less than -2 standard deviations
Infants' weight at birth (kg) | Birth
  Birth weight in kilograms using a seca scale, calculated as the mean of three repeated measurements on each infant
Percentage of infants with low birth weight | Birth
  Percentage of infants with birth weight less than 2500 grams
Percentage of preterm births | Birth
  Percentage of infants born with a gestational age less than 259 days
Percentage of infants who were small-for-gestational-age | Birth
  Percentage of infants at birth whose weight centiles were below the 10th percentile for their age and sex
Head circumference measurement (cm) | 0-2 years old
  Infant's head circumference measured in centimeters

SECONDARY OUTCOMES:
Percent of mothers that were anemic (hemoglobin levels <11 g/dL) | through study completion, every 3 months
  Percentage of maternal anemia defined by hemoglobin levels <11 g/dL, measured using the HemoCue test.
Percent of infants that were anemic (hemoglobin levels <11 g/dL) | 0-2 years old
  Percentage of infants with anemia defined by hemoglobin levels <11 g/dL, measured using the HemoCue test.
Concentration of ferritin (ug/L) in mothers and infants as a biomarker for iron status | 6 months for infants, mothers at birth
  Maternal and infants' serum ferritin (ug/L) measured using a sandwich enzyme-linked immunosorbent assay technique (ELISA) at the VitMin Lab in Germany
Concentration of soluble transferrin receptor (mg/L) in mothers and infants as a biomarker for iron status | 6 months for infants, mothers at birth
  Maternal and infants' serum soluble transferrin receptor (mg/L) measured using a sandwich enzyme-linked immunosorbent assay technique (ELISA) at the VitMin Lab in Germany
Concentration of retinol binding protein (umol/L) in mothers and infants as a biomarker for vitamin A status | 6 months for infants, mothers at birth
  Maternal and infants' serum retinol binding protein (umol/L) measured using a sandwich enzyme-linked immunosorbent assay technique (ELISA) at the VitMin Lab in Germany

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Webb, PhD, Study Director — Tufts, Friedman School of Nutrition; Shibani Ghosh, PhD, Principal Investigator — Tufts, Friedman School of Nutrition
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be publicly available by the end of 2020
Time Frame: End of 2020
Access Criteria: Data will be publicly accessible

REFERENCES:
- [Derived] Mezzano J, Namirembe G, Ausman LM, Marino-Costello E, Shrestha R, Erhardt J, Webb P, Ghosh S. Effects of Iron and Vitamin A Levels on Pregnant Women and Birth Outcomes: Complex Relationships Untangled Using a Birth Cohort Study in Uganda. Matern Child Health J. 2022 Jul;26(7):1516-1528. doi: 10.1007/s10995-022-03387-5. Epub 2022 Mar 3. PMID 35239084
- [Derived] Madzorera I, Ghosh S, Wang M, Fawzi W, Isanaka S, Hertzmark E, Namirembe G, Bashaasha B, Agaba E, Turyashemererwa F, Webb P, Duggan C. Prenatal dietary diversity may influence underweight in infants in a Ugandan birth-cohort. Matern Child Nutr. 2021 Jul;17(3):e13127. doi: 10.1111/mcn.13127. Epub 2021 Feb 17. PMID 33595899